CLINICAL TRIAL: NCT07389499
Title: A Clinical Study Evaluating the Safety and Efficacy of GT719 Universal Cell Injection in the Treatment of Immune-mediated Kidney Diseases
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRIT-CD-CHN-719-004-055
Record Dates: First submitted 2026-01-21; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: IgA Nephropathy (IgAN); Membranous Nephropathy; ANCA-associated Vasculitis (AAV)/ANCA-associated Glomerulonephritis (AAGN); Refractory Podocytopathy; Proliferative Glomerulonephritis With Monoclonal Immunoglobulin Deposits
MeSH Terms: conditions — Glomerulonephritis, IGA; Glomerulonephritis, Membranous; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GT719 Injection treatment group (Experimental): GT719 Injection
  Interventions: Biological: CD19-targeted iNKT Cell Injection

INTERVENTIONS:
Biological: CD19-targeted iNKT Cell Injection — Composed of CD19-targeted iNKT cells

SUMMARY:
This study is a single-arm, open-label, dose-escalation and dose-expansion clinical trial, divided into two phases: the first phase is the dose-escalation phase, and the second phase is the dose-expansion phase. In the dose-escalation phase, approximately 9-18 adult participants with immune-mediated kidney diseases are planned to be enrolled and treated with GT719 universal cell injection. The objectives of this phase are to evaluate the safety and tolerability of the product, determine the recommended dose (RD) for subsequent studies, conduct a preliminary assessment of its clinical efficacy, and investigate the pharmacokinetic and pharmacodynamic characteristics. Upon completion of the dose-escalation phase, after evaluation by investigators and collaborators, an appropriate dose will be selected for the dose-expansion phase. An additional 12 participants will be enrolled to fully assess the safety and efficacy of the product.

ELIGIBILITY:
Inclusion Criteria:

* 1. The participant or their legal representative voluntarily signs a written informed consent form, and is willing and able to comply with the procedures of this study.
* 2. Aged 18 to 75 years (inclusive) at the time of signing the informed consent, regardless of gender.
* 3. Positive expression of CD19 on B cells in peripheral blood is confirmed by flow cytometry.
* 4. Participants with IgA nephropathy (IgAN) at high risk of progression:

  ① A definite pathological diagnosis of IgAN confirmed by renal biopsy (renal biopsy must be performed within 2 years prior to screening or during the screening period).
  * Meet at least one of the following requirements:

    1. Prior treatment with glucocorticoids, budesonide enteric-coated capsules, immunosuppressants (including mycophenolate mofetil, cyclophosphamide, cyclosporine, tacrolimus, Tripterygium wilfordii, leflunomide, azathioprine), or biological agents (including but not limited to anti-CD20 monoclonal antibodies, telitacicept, daratumumab) for a cumulative duration of at least 3 months, with persistent 24-hour urinary protein ≥ 0.75 g or UPCR ≥ 0.75 g/g.
    2. The predicted probability of a 50% decline in eGFR or end-stage renal disease (ESRD) within 5 years calculated by the international IgAN prediction tool is ≥ 20%.
    3. A ≥ 20% decline in eGFR within 3 months.
    4. Renal biopsy performed within 6 months indicating Oxford classification C2 lesion.
    5. Patients who are intolerant to conventional treatment and for whom the investigator determines that the benefits outweigh the risks, with adequate informed consent obtained, may be considered for inclusion.
* 5. Participants with ANCA-associated vasculitis (AAV)/ANCA-associated glomerulonephritis (AAGN) must meet the following criteria:

  ① Diagnosis of granulomatosis with polyangiitis (GPA) or microscopic polyangiitis (MPA) according to the 2022 ACR/EULAR classification criteria for ANCA-associated vasculitis.

  ② Positive anti-myeloperoxidase (MPO-ANCA) antibody or anti-proteinase 3 (PR3-ANCA) antibody detected during screening or in previous tests.

  ③ AAGN: Availability of a renal biopsy pathological report within 2 years; if eGFR < 30 mL/min/1.73 m², a renal biopsy pathological report obtained during the screening period is required. Presence of active lesions according to the 2010 Berden classification criteria for AAGN.

  ④ Renal-uninvolved AAV: Birmingham Vasculitis Activity Score (BVAS) version 3.0 ≥ 3 points, indicating active vasculitis.

  ⑤ Failure of standard of care (SOC), defined as any of the following:

  a) Failure to achieve remission after at least 3 months of treatment with glucocorticoids combined with cyclophosphamide or rituximab.

  b) Disease relapse after achieving remission. c) Persistent disease activity despite receiving SOC for at least 6 months, including glucocorticoids, cyclophosphamide, rituximab, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, as well as other biological agents (including but not limited to mepolizumab) or avacopan.
* 6. Participants with membranous nephropathy (MN) must meet the following criteria:

  * Definite pathological diagnosis of primary (idiopathic) MN confirmed by renal biopsy (renal biopsy must be performed within 2 years prior to screening or during the screening period).

    ② Elevated serum anti-PLA2R antibody titer detected during screening or in previous tests, or positive PLA2R antigen staining in renal tissue.

    ③ eGFR ≥ 30 mL/min/1.73 m².

    ④ Meeting the criteria for high-risk or relapsed/refractory MN: c) High-risk patients, defined as meeting any of the following: Normal eGFR, urinary protein > 3.5 g/24h, < 50% reduction in urinary protein after 6 months of ACEI/ARB treatment, and serum albumin < 25 g/L or anti-PLA2R antibody > 50 RU/mL.

eGFR < 60 mL/min/1.73 m² and/or urinary protein > 8 g/24h for more than 6 months.

d) Relapsed/refractory patients: Relapsed patients: Defined as achieving complete or partial remission with previous SOC treatment, followed by recurrence of urinary protein ≥ 3.5 g/24h.

Refractory patients: Defined as refractory to previous SOC treatment (persistent urinary protein ≥ 3.5 g/24h with < 50% reduction compared to baseline).

* 7. Participants with refractory podocytopathy:

  ① Pathological diagnosis of minimal change disease (MCD) or focal segmental glomerulosclerosis (FSGS) confirmed by renal biopsy (renal biopsy must be performed within 2 years prior to screening or during the screening period).

  ② Meet at least one of the following requirements:
  1. Previous diagnosis of steroid-resistant nephrotic syndrome (SRNS): 24-hour urinary protein > 3 g or UPCR ≥ 3.5 g/g, serum albumin < 30 g/L, failure to achieve complete remission after 4 weeks of standard-dose glucocorticoid treatment.
  2. Previous diagnosis of steroid-dependent nephrotic syndrome (SDNS): Remission achievable with glucocorticoid treatment, but relapse within 2 weeks of glucocorticoid tapering or discontinuation, or two consecutive relapses during glucocorticoid tapering.
  3. Previous diagnosis of frequently relapsing nephrotic syndrome (FRNS): ≥ 3 relapses within 1 year or ≥ 2 relapses within 6 months after achieving complete remission with glucocorticoid treatment.
  4. Previous treatment with one immunosuppressant (including cyclosporine A, tacrolimus, mycophenolate mofetil, cyclophosphamide) or biological agent (including but not limited to anti-CD20 monoclonal antibodies, telitacicept, daratumumab) for ≥ 6 months without achieving remission or with intolerance.
  5. Failure to achieve remission within 6 months of adequate treatment with one immunosuppressant or biological agent, but the investigator judges that the benefits outweigh the risks and the patient has provided full informed consent, the patient may be considered for inclusion.
* 8. Participants with proliferative glomerulonephritis with monoclonal immunoglobulin deposition (PGNMID):

  * Definite pathological diagnosis of PGNMID confirmed by renal biopsy (renal biopsy must be performed within 3 years prior to screening or during the screening period).

    * Meet at least one of the following requirements:

Persistent 24-hour urinary protein ≥ 1 g or UPCR ≥ 1 g/g despite treatment with angiotensin-converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) for at least 4 weeks.

eGFR ≥ 30 mL/min/1.73 m² with progressive decline (≥ 20% decrease in eGFR) within the recent 6-12 months.

Development of nephrotic syndrome or nephrotic-range proteinuria (24-hour urinary protein ≥ 3 g or UPCR ≥ 3 g/g) without stable remission with short-term glucocorticoid treatment.

③ Exclusion of hematological malignancies (leukemia, lymphoma, multiple myeloma, systemic light chain amyloidosis) by bone marrow aspiration and biopsy (bone marrow aspiration must be performed within 6 months prior to screening or during the screening period).

* 9. Screening laboratory test results must meet the following criteria (excluding indicators related to the study disease):

  1. Neutrophil count ≥ 1.5 × 10⁹/L;
  2. Hemoglobin ≥ 80 g/L; Platelet count ≥ 50 × 10⁹/L;
  3. Alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN); Aspartate aminotransferase (AST) ≤ 3 × ULN; Total bilirubin (TBIL) < 2 × ULN (for participants with Gilbert syndrome, direct bilirubin (DBIL) ≤ 1.5 × ULN);
  4. Creatinine clearance rate ≥ 30 mL/min; (except for anti-GBM glomerulonephritis, AAV/ANCA-associated glomerulonephritis);
  5. Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; Prothrombin time (PT) ≤ 1.5 × ULN;
  6. Left ventricular ejection fraction (LVEF) ≥ 50% diagnosed by echocardiography.
  7. Pulmonary function: Defined as dyspnea ≤ CTCAE Grade 1 and oxygen saturation (SpO₂) ≥ 92% at rest while breathing room air (measured by pulse oximetry).
* 10. Female participants of childbearing potential must:

  a. Have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result at screening, confirmed by the investigator; b. Agree to avoid breastfeeding during study participation until at least 1 year after GT719 cell infusion or until GT719 cells are no longer detected by two consecutive flow cytometry tests, whichever is later.
* 11. Male participants with sexual partners and female participants of childbearing potential must agree to use highly effective contraceptive methods (e.g., contraceptive pills, intrauterine devices, or condoms) starting from screening until at least 1 year after GT719 cell infusion or until GT719 cells are no longer detected by two consecutive flow cytometry tests, whichever is later. Male participants must agree to use condoms during sexual contact with pregnant women or women of childbearing potential for at least 1 year after GT719 cell infusion, even after successful vasectomy.

Exclusion Criteria:

* 1. Participants with IgA nephropathy (IgAN) at high risk of progression:

  a. Secondary IgAN (e.g., associated with active hepatitis B/hepatitis C infection, HIV, etc.).
* 2. Participants with ANCA-associated vasculitis (AAV)/ANCA-associated glomerulonephritis (AAGN):

  1. Drug-induced or secondary AAV/AAGN.
  2. Alveolar hemorrhage requiring invasive mechanical ventilation support at screening.
* 3. Participants with membranous nephropathy (MN):

  a. Secondary membranous nephropathy.
* 4. Participants with refractory podocytopathy:

  a. Hereditary podocytopathy and secondary focal segmental glomerulosclerosis (FSGS).
* 5. Participants with proliferative glomerulonephritis with monoclonal immunoglobulin deposition (PGNMID):

  1. Monoclonal deposition caused by secondary nephropathy (e.g., those diagnosed with multiple myeloma or severe systemic lymphoplasmacytic disease requiring immediate oncological treatment).

For all participants:

* 6. History of severe hypersensitivity reaction or allergy.
* 7. Contraindication or hypersensitivity to fludarabine, cyclophosphamide, or any component of the investigational product.
* 8. Currently receiving renal replacement therapy or expected to require renal replacement therapy during the study period.
* 9. Rapidly progressive glomerulonephritis unrelated to AAV/AAGN, anti-GBM disease, MN, acute post-streptococcal nephritis (APSN), or IgG4-related kidney disease (IgG4-RKD), defined as a ≥ 50% decrease in eGFR within 3 months of diagnosis.
* 10. History of other uncontrolled severe conditions not directly related to the study disease prior to screening, such as severe hemolytic anemia, severe immune thrombocytopenic purpura, severe agranulocytosis, severe myocardial damage, severe pneumonia or pulmonary hemorrhage, severe hepatitis, severe vasculitis, active central nervous system (CNS) symptoms including cerebrovascular accident, aneurysm, epilepsy, convulsion, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis.
* 11. History of the following cardiac diseases or conditions:

  1. New York Heart Association (NYHA) Class III or IV congestive heart failure within 12 months prior to screening;
  2. Myocardial infarction or coronary artery bypass grafting within 6 months prior to screening;
  3. History of clinically significant ventricular arrhythmia or unexplained syncope not caused by vasovagal response or dehydration, or corrected QT interval (QTc) > 480 ms at screening;
  4. History of severe non-ischemic cardiomyopathy;
  5. Pulmonary arterial hypertension, including secondary pulmonary arterial hypertension, with WHO functional class > 2;
  6. QTcF > 450 msec in males and QTcF > 470 msec in females, based on the average QTcF (QT interval corrected by Fridericia's formula) value from a single ECG or three repeated ECGs performed at intervals of more than 3 minutes.
* 12. Presence of significant pulmonary or cardiac manifestations (e.g., pericarditis, pleural effusion) at screening, which the investigator assesses may affect the participant's ability to receive treatment safely or tolerate treatment.
* 13. Evidence of advanced fibrotic interstitial lung disease on chest CT, with the latest pulmonary function test showing forced vital capacity (FVC) < 40% of predicted value or diffusing capacity of the lung for carbon monoxide (DLCO) < 30% of predicted value.
* 14. History of any active malignancy or malignant tumor within 5 years prior to screening. Exceptions include: early-stage tumors treated with radical therapy (carcinoma in situ or Stage I tumor, non-ulcerative primary melanoma with depth < 1 mm and no lymph node involvement), cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, cervical carcinoma in situ, or ductal carcinoma in situ of the breast that has received potentially curative treatment.
* 15. Clinically significant bleeding symptoms or definite bleeding tendency within 6 months prior to screening, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, etc.; hereditary or acquired bleeding and thrombotic tendency (e.g., hemophilia, coagulation dysfunction, hypersplenism, etc.); occurrence of arteriovenous thrombotic events within 6 months prior to screening, such as cerebrovascular disease (including cerebral hemorrhage, cerebral infarction, etc.), deep vein thrombosis, and/or pulmonary embolism.
* 16. Presence of severe underlying medical conditions at screening, such as:

  1. Evidence of uncontrolled viral, bacterial, fungal, or other infections requiring systemic intravenous treatment;
  2. Obvious clinical evidence of dementia or altered mental status;
  3. History of any other CNS disease or neurodegenerative disease, such as epilepsy, convulsion, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, or psychosis.
* 17. Positive results for any of the following tests:

  1. Human immunodeficiency virus (HIV) antibody positive;
  2. Hepatitis B surface antigen (HBsAg) positive; or hepatitis B core antibody (HBcAb) positive with hepatitis B virus (HBV)-DNA level above the lower limit of quantification (LLOQ) of the assay;
  3. Hepatitis C virus (HCV) antibody positive with HCV RNA level above the LLOQ of the assay;
  4. Syphilis antibody positive (excluding false-positive results caused by underlying diseases).
* 18. H Positive results for cytomegalovirus (CMV) DNA or Epstein-Barr virus (EBV) DNA test.
* 19. Active tuberculosis prior to screening or latent tuberculosis not receiving appropriate treatment.
* 20. Receipt of other investigational drugs within 4 weeks prior to signing the informed consent form (ICF), or the interval between the ICF signing date and the last dose of the previous investigational drug trial is still within 5 half-lives of the drug, whichever is longer.
* 21. Receipt of plasma exchange therapy or immunoadsorption therapy within 4 weeks prior to lymphodepletion conditioning.
* 22. Receipt of B-cell-targeted drug therapy within 1 week prior to lymphodepletion conditioning, including but not limited to rituximab, obinutuzumab, belimumab, telitacicept, etc.
* 23. Receipt of tacrolimus, cyclosporine, azathioprine, mycophenolate mofetil, mycophenolic acid, methotrexate, etc., within 2 weeks prior to lymphodepletion conditioning.
* 24. Receipt of neonatal Fc receptor (FcRn) antagonist therapy (e.g., efgartigimod, etc.) within 3 weeks prior to lymphodepletion conditioning.
* 25. Receipt of complement inhibition therapy (e.g., eculizumab, etc.) within 3 weeks prior to lymphodepletion conditioning.
* 26. Receipt of live attenuated vaccine within 4 weeks prior to lymphodepletion conditioning.
* 27. Performance of major surgery within 8 weeks prior to screening, or planned surgery during the study period.
* 28. History of organ transplantation.
* 29. Previous receipt of CAR-T product therapy targeting any antigen (except for GT719 treatment).
* 30. Presence of any condition that, in the investigator's judgment, would prevent the participant from completing the entire trial, confound trial results, or make trial participation not in the participant's best interest.
* 31. Presence of donor-specific anti-HLA antibodies against GT719 cells.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability: Evaluate the incidence, correlation with the investigational product, severity, and other relevant aspects of adverse events (AEs) and serious adverse events (SAEs) occurring in participants during the trial | 24 Months
  Based on the current version of the Common Terminology Criteria for Adverse Events (CTCAE) developed by the National Cancer Institute (NCI) of the United States, a systematic assessment of the safety and tolerability of the study subjects was conducted throughout the entire trial period.
Changes in vital signs before and after treatment | 1 Month
  Dynamic monitoring of changes in vital signs before and after treatment, including heart rate, body temperature, blood pressure, etc.
Changes in clinical symptoms before and after treatment | 1 Month
  A comparative analysis of the dynamic changes in clinical symptoms before and after treatment, including skin changes, pulmonary conditions, etc., is planned to be conducted.
Changes in laboratory tests before and after treatment | 1 Month
  A comparative analysis of the dynamic changes in laboratory test indicators, including blood routine, blood biochemistry, relevant antibodies, etc., is planned to be conducted.
Changes in electrocardiograms before and after treatment | 1 Month
  A comparative analysis of the dynamic changes in electrocardiograms is planned to be conducted.

SECONDARY OUTCOMES:
All Participants: Time to Maximum Expansion of Infused Cells (Tmax) | 24 Months
  The time point at which the concentration of infused cells in peripheral blood reaches the peak level following product infusion, measured by flow cytometry.
All Participants: Peak Expansion Level of Infused Cells (Cmax) | 24 Months
  The maximum copy number or cell count of infused cells in peripheral blood after infusion, measured by flow cytometry.
All Participants: Area Under the Curve of Infused Cells (AUC) | 24 Months
  The area under the concentration-time curve of infused cells in peripheral blood from the time of infusion to the evaluation endpoint, reflecting the total exposure of cells in vivo.
All Participants: Duration of Observable Concentration (Tlast) | 24 Months
  The time period during which the concentration of a drug, cell (e.g., CAR-T cell), or biomarker in the body can be stably detected continuously after reaching or exceeding the Lower Limit of Quantitation (LLOQ) of the detection method.
All Participants: CAR-T-associated Serum Cytokines | 2 Months
  A class of soluble protein molecules whose release or expression levels in patients' serum undergo significant changes due to the activation, proliferation of CAR-T cells or their interaction with target cells after CAR-T cells are infused into patients' bodies.
All Participants: CAR Cell Phenotype | 24 Months
  The inherent biological properties exhibited by T cells expressing chimeric antigen receptors (CARs) (i.e., CAR-T cells) in terms of morphology, surface marker expression, and functional characteristics.
Participants with IgA nephropathy at high risk of progression：The proportion of participants who achieved complete response and partial response at 28 days, as well as at Months 2, 3, 6 and 12. | Day 28, Month 2, 3, 6 and 12
  The remission status of the subjects was statistically analyzed at five key time points: 28 days, 2 months, 3 months, 6 months, and 12 months after treatment. The proportions of subjects who achieved complete response (CR) and partial response (PR) at each time point relative to the total enrolled subjects were calculated.
Participants with IgA nephropathy at high risk of progression： The estimated glomerular filtration rate (eGFR) slope at Day 14, Day 28, Month 2, Month 3, Month 6, and Month 12 | Day 14 and 28, Month 2, 3, 6, and 12
  Using estimated glomerular filtration rate (eGFR) as the core indicator for evaluating the dynamic changes in renal function, the eGFR slopes of the subjects were calculated separately at six key time points: 14 days, 28 days, 2 months, 3 months, 6 months, and 12 months after treatment.
Participants with ANCA-Associated Vasculitis (AAV)/ANCA-Associated Glomerulonephritis (AAGN): The proportion of participants who achieved complete response (CR) and partial response (PR) at 28 days, as well as at Months 2, 3, 6, and 12 | Day 28, Month 2, 3, 6 and 12
  The remission status of the subjects was statistically analyzed at five key time points: 28 days, 2 months, 3 months, 6 months, and 12 months after treatment. The proportions of subjects who achieved complete response (CR) and partial response (PR) at each time point relative to the total enrolled subjects were calculated.
Participants with ANCA-Associated Vasculitis (AAV)/ANCA-Associated Glomerulonephritis (AAGN): Changes in ANCA-MPO or PR3 antibody levels relative to baseline at Day 14, Day 28, as well as at Months 2, 3, 6, and 12 | Day 14 and 28, Month 2, 3, 6, and 12
  With anti-neutrophil cytoplasmic antibody-myeloperoxidase (ANCA-MPO) and anti-neutrophil cytoplasmic antibody-proteinase 3 (ANCA-PR3) as the core detection indicators, blood samples were collected from the subjects at baseline before treatment, as well as at Day 14, Day 28, Month 2, Month 3, Month 6, and Month 12 after treatment, and a standardized detection method was used for the quantitative determination of antibody levels.
Participants with ANCA-Associated Vasculitis (AAV)/ANCA-Associated Glomerulonephritis (AAGN): Changes in Birmingham Vasculitis Activity Score (BVAS) relative to baseline at 28 days, as well as at Months 2, 3, and 6 | Day 28, Month 2, 3 and 6
  With the Birmingham Vasculitis Activity Score (BVAS) as the core assessment tool for vasculitis disease activity, standardized scoring of the subjects was performed by uniformly trained evaluators at five time points: baseline before treatment, 28 days, 2 months, 3 months, and 6 months after treatment.
Participants with Membranous Nephropathy (MN): The proportion of participants who achieved complete response (CR) and partial response (PR) at 28 days, as well as at Months 2, 3, 6, and 12 | Day 28, Month 2, 3, 6 and 12
  The remission status of the subjects was statistically analyzed at five key time points: 28 days, 2 months, 3 months, 6 months, and 12 months after treatment. The proportions of subjects who achieved complete response (CR) and partial response (PR) at each time point relative to the total enrolled subjects were calculated.
Participants with Membranous Nephropathy (MN) : Changes in anti-PLA₂R antibody levels relative to baseline at Day 14, Day 28, as well as at Months 2, 3, 6, and 12 | Day 14 and 28, Month 2, 3, 6, and 12
  Using anti-phospholipase A₂ receptor antibody (anti-PLA₂R antibody) as the core biomarker for evaluating the disease activity and treatment response of membranous nephropathy, peripheral blood samples were collected from the subjects at seven key time points: baseline before treatment, Day 14, Day 28, Month 2, Month 3, Month 6, and Month 12 after treatment.
Participants with refractory podocytopathy: The proportion of participants who achieved complete response (CR) and partial response (PR) at 28 days, as well as at Months 2, 3, 6, and 12 | Day 28, Month 2, 3, 6 and 12
  The remission status of the subjects was statistically analyzed at five key time points: 28 days, 2 months, 3 months, 6 months, and 12 months after treatment. The proportions of subjects who achieved complete response (CR) and partial response (PR) at each time point relative to the total enrolled subjects were calculated.
Participants with refractory podocytopathy: The recurrence rate of nephrotic syndrome within 12 months | 12 Months
  With the recurrence of nephrotic syndrome as the key evaluation endpoint, the recurrence status of the subjects was statistically analyzed during the 12-month follow-up period after the first achievement of remission (complete response/partial response).
Proliferative Glomerulonephritis with Monoclonal Immunoglobulin Deposits (PGNMID): The proportion of participants who achieved complete response (CR) and partial response (PR) at 28 days, as well as at Months 2, 3, 6, and 12 | Day 28, Month 2, 3, 6 and 12
  The remission status of the subjects was statistically analyzed at five key time points: 28 days, 2 months, 3 months, 6 months, and 12 months after treatment. The proportions of subjects who achieved complete response (CR) and partial response (PR) at each time point relative to the total enrolled subjects were calculated.
PGNMID: The proportion of participants with normalization of serum free light chain ratio (for those with abnormal baseline levels), and the negative rate of serum/urine immunofixation electrophoresis at Day 14, Day 28, as well as at Months 2, 3, 6, 12 | Day 14 and 28, Month 2, 3, 6, and 12
  Peripheral blood and urine samples were collected from the subjects at seven key time points: baseline before treatment, Day 14, Day 28, Month 2, Month 3, Month 6, and Month 12 after treatment. The serum free light chain κ/λ ratio was determined by immunoturbidimetry, and monoclonal immunoglobulin bands in blood and urine samples were identified by immunofixation electrophoresis.

OTHER OUTCOMES:
Peripheral Blood Lymphocyte Subsets | 24 Months
  Lymphocyte populations in peripheral blood with distinct surface markers and functional characteristics.
Exploration of T Cells by B Lymphocyte Subsets | 24 Months
  Taking B lymphocyte subsets as the research tool/entry point, this study explores their interaction with T cells, as well as the functional impacts and regulatory mechanisms involved.
Changes in NK cells | 24 Months
  Detect the dynamic changes in the quantity, proportion, activity, and phenotypic characteristics of natural killer (NK) cells.
HLA Typing/Antibody Changes | 28 days after informed consent
  The dynamic changes in the genotyping characteristics of Human Leukocyte Antigen (HLA) and the anti-HLA antibody profile in the body.
Duration of B Cell Depletion | 24 Months
  The time span during which the number of B cells in the peripheral blood or tissues of the body drops below the baseline level and remains at a low level after immune intervention.
Explore and analyze the diversity of the BCR repertoire by means of BCR sequencing | 24 Months
  BCR repertoire diversity refers to the richness of the gene sequences, clonal types, and variable region (V-D-J) recombination patterns of B cell receptors in the body, and its diversity level directly reflects the body's potential for immune responses against antigen stimulation.
Pathological Changes of Affected Organs Before and After Treatment | 24 Months
  The dynamic changes in the histological morphology, cellular phenotype, degree of inflammatory infiltration, and injury repair status of target organs damaged during disease progression, before and after interventions such as medication, cellular therapy, and surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No